CLINICAL TRIAL: NCT02346890
Title: A Phase 1, Single-center, Randomized, 2-way Crossover, Open Label Study to Evaluate the Effect of Renvela on the Pharmacodynamics of AZD1722 in Healthy Volunteeers
Brief Title: A Phase 1 Study to Examine the Effect of Renvela on the Pharmacodynamics of AZD1722
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5611C00006
Record Dates: First submitted 2014-09-24; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Volunteer
MeSH Terms: interventions — tenapanor; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1722 alone (Experimental): 15 mg BID
  Interventions: Drug: AZD1722
- AD1722 with Renvela (Experimental): AZD1722 15 mg BID and Renvela 800 mg TID
  Interventions: Drug: AZD1722; Drug: Renvela

INTERVENTIONS:
Drug: AZD1722
  Other Names: RDX5791; Tenapanor
Drug: Renvela
  Other Names: Sevelamer carbonate
  Arms: AD1722 with Renvela

SUMMARY:
The study is designed to evaluate safety, tolerability, pharmacodynamics and pharmacokinetics of AZD1722 in healthy volunteers taking Renvela.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman
* Body mass index between 18 and 29.9 kg/m2

Exclusion Criteria:

* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the gastrointestinal (GI) tract
* Any surgery on the small intestine or colon, excluding appendectomy or cholecystectomy or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, metabolic, endocrine, neurologic, psychiatric disease, or any condition that may interfere with the subject successfully completing the trial or that would present a safety risk to the subject.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Sodium levels in stool and urine | 4 days
  Pharmacodynamic activity

SECONDARY OUTCOMES:
Evaluate the safety of AZD1722, measured by Adverse events | 8 days
  Adverse events
Evaluate the safety of AZD1722, measured by clinical laboratory changes | 8 days
  clinical laboratory changes
Plasma drug concentration to calculate AUC | 8 days
  Evaluate the Pharmacokinetics of AZD1722

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Director — Ardelyx, Inc.
Locations (1):
- Healthcare Discoveries, LLC, San Antonio, Texas, United States